CLINICAL TRIAL: NCT05575557
Title: Pulmonary Artery Pressure and Right Heart Evaluation for Patients Requiring Physiological Pacing Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, Head of Cardiology, Shanghai 10th People's Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PROPHET
Record Dates: First submitted 2022-09-17; First posted 2022-10-12 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-10

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Atrial Fibrillation, Persistent; Sick Sinus Syndrome; Atrioventricular Block
Keywords: physiological pacing; right heart; hemodynamics examination; acute and chronic impact
MeSH Terms: conditions — Atrial Fibrillation; Sick Sinus Syndrome; Atrioventricular Block

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- His bundle pacing group (Active Comparator): HBP was performed on the patient, and the detection of the His bundle potential during the procedure is the sign of the success of the procedure. The HB capture threshold was accepted if lower than 3.0 V at 0.42ms.
  Interventions: Procedure: Right heart catheterization
- Left branch bundle pacing group (Active Comparator): HBP was performed on the patient, and the detection of the His bundle potential during the procedure is the sign of the success of the procedure. During the procedure, the duration from the pacing signal to the peak of R wave (on V4-V6 lead) is measured as pacing to left ventricular activation time (p-LVAT). An eligible site of left bundle capture was confirmed if selective LBBP was demonstrated by ECG, if p-LVAT shortened abruptly >10 ms through increasing pacing output, or if p-LVAT stayed shortest and stable at the site.
  Interventions: Procedure: Right heart catheterization
- Right ventricular pacing group (Active Comparator): If we could not achieve an acceptable HB or LBB capture after five attempts of lead positioning or a fluoroscopy exposure time over 30min, the lead was then placed in the RV with traditional approach.
  Interventions: Procedure: Right heart catheterization

INTERVENTIONS:
Procedure: Right heart catheterization — All groups were detected with SW catheter by the internal jugular vein before the procedure. After the measurement, the catheter was indwelled, and the pacemaker implantation procedure was started. After ventricular pacing for 5 minutes, the SW catheter measurement was performed again. After the measurement, the SW catheter was withdrawn.

SUMMARY:
With the aging of society, the use of cardiac pacing in patients with irreversible bradycardia is increasingly widespread. As early as the 1950s, right ventricular pacing (RVP) began to be used in patients with atrioventricular block or sick sinus syndrome, but in fact such pacing could cause ventricular asynchrony, which could lead to long-term myocardial perfusion injury, valvular regurgitation, heart failure, and increased risk of ventricular tachycardia and ventricular fibrillation. The latest guideline recommended reducing the proportion of right ventricular pacing. Additionally, in patients with heart failure with reduced ejection fraction (EF ≤ 35%) and complete left bundle branch block, cardiac resynchronization therapy (CRT) with biventricular pacing (BVP) has been recommended to improve cardiac function, but only about 30% of patients benefit from it, which may be related to poor left ventricular pacing site and myocardial scarring. In theory, His bundle pacing (HBP) compared with RVP can reduce the risk of functional tricuspid regurgitation when the lead position lies on the atrial side of the tricuspid valve, which may improve the right heart function and pulmonary artery pressure. In 2021, Domenico Grieco et al. explored the effect of HBP on right heart function. After 6 months of follow-up, it was found that HBP improved right heart function and pulmonary artery pressure compared with RVP.

At present, there are few discussions on the effect of physiological pacing on right ventricular hemodynamics, and the sample size is small. Internationally, the discussion of the assessment of hemodynamics is limited to non-invasive evaluation (such as echocardiography, ECG, SPECT) The gold standard for right heart hemodynamics evaluation is the measurement of invasive right heart catheterization, and there has been no relevant research so far, so the investigators further designed a study of the effect of physiological pacing on hemodynamics.

DETAILED DESCRIPTION:
This study was designed to investigate the acute and chronic effect of different pacing methods on the function of pulmonary artery and right heart.

Studied population: The investigated population are patients eligible for pacemaker implantation and cardiac resynchronization therapy and specified as followed:

1. age over 18; 2. persistent atrial fibrillation patients with uncontrolled heart rate requiring atrioventricular node ablation; 3. heart failure patients with EF≤35% and complete left bundle branch block; 4. patients with sick sinus syndrome or atrioventricular block eligible for pacemaker implantation.

Investigated procedure: Physiological pacing as the principal studied procedure is defined as pacing with ventricular lead implanted at proximal/distal His bundle or left bundle branch. While right ventricular pacing was defined as conventional pacing with ventricular lead implanted at right ventricular apex.

Importantly, Swan-Ganz catheter was performed before and after physiological pacing. By the internal jugular vein before the pacemaker implantation procedure. After the measurement, the catheter was indwelled and measurement was taken. Thereafter, pacemaker implantation procedure was followed. After completing electrode fixation and continuous ventricular pacing for at least 5 minutes, ensuring ventricular pacing ratio > 80%, the SW catheter measurement was performed again to acquire indices under physiological pacing.

Follow up: The study is designed to have scheduled follow-up at 1 month, 3-month, 6-month and 12 months after procedure. Primary endpoint is a composite endpoint of all-cause mortality and HF rehospitalization. And other imageological measurement (echocardiography) biochemical test (blood BNP) and functional evaluation (6MWT) were performed to appraise the impact of physiological pacing on the condition of the participants.

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* persistent atrial fibrillation patients with uncontrolled heart rate requiring atrioventricular node ablation
* patients with sick sinus syndrome or atrioventricular block eligible for pacemaker implantation
* patients who can understand and sign informed consent

Exclusion Criteria:

* age below 18 or over 99
* concomitant diseases that may affect right heart function, including COPD, pulmonary infection, history of pulmonary embolism or right myocardial infarction, myocarditis, systemic disease
* patients with temporary pacemaker implanted
* right heart catheterization contraindications, including acute infection and embolic events

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events after procedure | From date of inclusion until the date of documented adverse events, assessed up to 1 year
  rehospitalization due to acute heart failure, all-cause mortality, cardiac death

SECONDARY OUTCOMES:
Changes in systolic, diastolic and mean pulmonary artery pressure by Swan-Ganz catheter from pre-procedure level | 5 minutes after ventricular pacing lead implantation
  Measurement of systolic, diastolic and pulmonary artery pressure by Swan-Ganz catheter before and 5 minutes after ventricular pacing lead implantation
Changes in systolic, diastolic and mean right ventricular pressure by Swan-Ganz catheter from pre-procedure level | 5 minutes after ventricular pacing lead implantation
  Measurement of systolic, diastolic and mean right ventricular pressure by Swan-Ganz catheter before and 5 minutes after ventricular pacing lead implantation
Changes in systolic, diastolic and mean right atrial pressure by Swan-Ganz catheter from pre-procedure level | 5 minutes after ventricular pacing lead implantation
  Measurement of systolic, diastolic and mean right atrial pressure by Swan-Ganz catheter before and 5 minutes after ventricular pacing lead implantation
Changes in right ventricular global longitudinal strain rate from pre-porcedure level | 24 hours post procedure, 1st month, 3rd month, 12th month since procedure
  Right ventricular global longitudinal strain rate measured at four-chamber view
Changes in tricuspid annular plane systolic excursion from pre-procedure level | 24 hours post procedure, 1st month, 3rd month, 12th month since procedure
  Tricuspid annular plane systolic excursion by tissue doppler imaging measured at four-chamber view
Changes in Tei index from pre-procedure level | 24 hours post procedure, 1st month, 3rd month, 12th month since procedure
  Tei index calculated from measurement by tissue doppler imaging of tricuspid moving velocity at four-chamber view
Changes in pulmonary artery systolic pressure by echocardiography from pre-procedure level | 24 hours post procedure, 1st month, 3rd month, 12th month since procedure
  Pulmonary artery systolic pressure was approximated by echocardiography measuring tricuspid regurgitation pressure
Change from baseline walking distance of 6-min walk test between different groups at 6 month after procedure | 1st month, 3rd month, 12th month since procedure
  Maximum walking distance measured from 6-min walk test
Change from baseline general quality of life evaluation | 1st month, 3rd month, 12th month since procedure
  Change in EQ-5D-5L questionnaire score
Change from baseline heart failure-specific quality of life evaluation | 1st month, 3rd month, 12th month since procedure
  Change in Kansas City Cardiomyopathy Questionnaire score
Change in heart failure biomarker from baseline | 1st month, 3rd month, 12th month since procedure
  Change in level of blood brain natriuretic peptide
Changes in blood pressure from baseline between different groups at 6 months after procedure | 1st month, 3rd month, 12th month since procedure
  Change of systolic and diastolic blood pressure, an average value of three times

CONTACTS AND LOCATIONS:
Overall Officials: Yawei Xu, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China